CLINICAL TRIAL: NCT07376629
Title: A Phase II Study of HB0025 in Combination With Nab-Paclitaxel as First Line Therapy for Unresectable, Locally Advanced or Metastatic Triple-negative Breast Cancer.
Brief Title: A Study of HB0025 Plus Nab-paclitaxel as First Line Therapy for TNBC
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB0025-C-0201
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: TNBC
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB0025 20mg/kg (Experimental)
  Interventions: Drug: HB0025 20 mg/kg plus nab-paclitaxel
- HB0025 10mg/kg (Experimental)
  Interventions: Drug: HB0025 10 mg/kg plus nab-paclitaxel

INTERVENTIONS:
Drug: HB0025 20 mg/kg plus nab-paclitaxel — HB0025 20 mg/kg
  Arms: HB0025 20mg/kg
Drug: HB0025 10 mg/kg plus nab-paclitaxel — HB0025 10 mg/kg
  Arms: HB0025 10mg/kg

SUMMARY:
This trial is a Phase II study. The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of HB0025 administered with chemotherapy in participants with locally advanced or metastatic triple-negative breast cancer (TNBC) who have not received prior systemic therapy for metastatic breast cancer (mBC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
3. No prior systemic therapy for inoperable locally advanced or metastatic TNBC
4. ECOG performance status of 0 or 1
5. Life expectancy ≥ 12 weeks
6. Measurable disease, as defined by RECIST v1.1

Exclusion Criteria:

1. History of severe allergic diseases, allergic history of serious drugs (including unlisted test drugs) or known allergic to any component of this test drug;
2. Previously received any antibody or inhibitor therapy targeting PD-1/PD-L1 or VEGF;
3. Uncontrollable or symptomatic central nervous system (CNS) metastasis;
4. Pregnancy or lactation;
5. Those who have active infection
6. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability measures: Incidence,correlation, and severity of adverse events graded according to NCI CTCAE v5.0. | From first dose to the time of the disease progression, intolerable toxicity, initiation of new antitumor therapy, loss to follow-up, death, withdrawal of study, completion of 2-year treatment of HB0025, or other reasons, whichever comes first.
  Safety profile including adverse events, changes in safety assessment parameters. Incidence, severity, outcome, and correlation to the study drug of all adverse events (AE), treatment-emergent adverse events (TEAE), serious adverse events (SAE) and adverse events of special interest (AESI) assessed according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0; Changes in vital signs, ECOG score, physical examination, electrocardiogram, and laboratory test results before and after study treatment.

SECONDARY OUTCOMES:
ORR per RECIST 1.1 for Part B | Week 3
  From first dose to the time of the disease progression, intolerable toxicity, initiation of new antitumor therapy, loss to follow-up, death, withdrawal of study, completion of 2-year treatment of HB0025, or other reasons, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Anyang Cancer Hospital, Anyang
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Fujian Cancer Hospital, Fujian
  - Guangdong Provincial People's Hospital, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - The First Hospital of Jilin University, Jilin
  - Affiliated Hospital of Jining Medical University, Jining
  - Linyi Cancer Hospital, Linyi
  - Jiangsu Province Hospital, Nanjing
  - Shandong Cancer Hospital, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanxi Cancer Hospital, Shanxi
  - Liaoning Cancer Hospital, Shengyang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Cancer Hospital, Tianjing
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xuzhou Central Hospital, Xuzhou

IPD SHARING:
Plan to Share IPD: Undecided
n